CLINICAL TRIAL: NCT05118685
Title: A Comparative Study of Vaginal Oestrogen Cream and Platelet Rich Plasma in Treatment of Atrophic Vaginitis in Fayoum University Hospital
Brief Title: Estrogen and Platelet Rich Plasma in Treatment of Atrophic Vaginitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, rehab abdelhamid aboshama, lecturer of obstetrics and gynecology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R 180
Record Dates: First submitted 2021-09-29; First posted 2021-11-12 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Atrophic Vaginitis; Postmenopausal Atrophic Vaginitis
Keywords: atrophic vaginitis; Platelet rich plasma; postmenopausal symptoms
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial that will be performed in a Fayoum university hospital. It includes 100 pt. complaining of atrophic vaginitis it will be divided into two groups, each group will contain 50 pt
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the first group estrogen group (Active Comparator): they will receive estrogen conjugate vaginal cream one tube every night for 14 nights; then, one tube 2 nights in 1 week (two tubes every week) for 10 weeks.
  Interventions: Drug: Conjugated Estrogens vaginal cream 0,625mg
- the second group PRP group (Experimental): they will receive a Platelet-rich plasma injection every 3 weeks for 4 times. PRP will be administered to the anterior vaginal wall using 27-G needles o and it is mainly injected into the anterior wall of the vagina to increase the tactile sensitivity of the injection site.
  Interventions: Combination Product: platelet rich plasma

INTERVENTIONS:
Drug: Conjugated Estrogens vaginal cream 0,625mg — the particepant will receive vaginal estrogen cream one tube every night for 14 nights; then, one tube for 2 nights in 1 week (two tubes every week) for 10 weeks.
  Other Names: Premarin cream
  Arms: the first group estrogen group
Combination Product: platelet rich plasma — First, a topical anesthetic cream will be applied to the vaginal wall. Delaying the PRP injection for 20 minutes after anesthetics application achieved complete or near-complete analgesia for the procedure. Peripheral blood will be drawn from the arm and centrifuged to yield 5 cc of PRP. then PRP will be administered to the anterior vaginal wall using 27-G needles once every 3 weeks for 4 times and PRP is mainly injected into the anterior wall of the vagina to increase the tactile sensitivity of the injection site.
  Arms: the second group PRP group

SUMMARY:
This study is designed to compare the efficacy, acceptability, and safety of vaginal estrogen cream and platelet-rich plasma in pt. complaining of atrophic vaginitis.

DETAILED DESCRIPTION:
Oestrogen deficiency affects many organs such as the genitourinary system. Genitourinary involvement causes untoward symptoms of atrophic vaginitis including dryness, burning, dyspareunia, vulvar pruritus, and discharge For this reason, many investigations have been performed to find out effective, safe, and acceptable therapeutic methods for atrophic vaginitis. Although systemic administration of estrogen can improve the localized symptoms of atrophic vaginitis, women are often reluctant to use systemic hormone replacement therapy and prefer local administration of estrogen. Vaginal application of estrogen has been considered an effective treatment of atrophic vaginitis.

The effects of PRP treatment have been evaluated in many clinical conditions, including wound healing, hair repair, skin regeneration [9], vulvar lichen sclerosis, stress urinary incontinence, episiotomy scars, and lubrication aging in the vagina. It can take at least 12 weeks to determine the final effects of treatment with PRP Population of Study It includes 100 pt. complaining of atrophic vaginitis it will be divided into two groups, each group will contain 50 pt

Methodology in detail:

Patients of the first group will receive vaginal estrogen cream one tube every night for 14 nights; then, one tube 2 nights in 1 week (two tubes every week) for 10 weeks.

The second group will receive PRP injection every 3 weeks for 4 times. PRP will be administered to the anterior vaginal wall using 27-G needles once every 3 weeks for 4 times and PRP is mainly injected into the clitoris or the anterior wall of the vagina to increase the tactile sensitivity of the injection site.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women aged 50-70 years old
* with a clinical diagnosis of vaginal atrophy who will not need systemic estrogen therapy for the treatment of vasomotor symptoms or prophylaxis of osteoporosis
* Any parity.

Exclusion Criteria:

* Women with any history of carcinoma of the breast or endometrium,
* abnormal genital bleeding, acute thrombophlebitis, or thromboembolic disorders associated with previous estrogen use,
* or current urinary.
* In addition, women who underwent hormone replacement therapy, treated with systemic or vaginal estrogen within 6 months prior to the study,
* or had any contraindication for estrogen therapy will be excluded from the study.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal atrophic vaginitis
Enrollment: 100 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
improvement in Vaginal Health Index (VHI). | 12 weeks
  Vaginal Health Index (VHI) will be assessed at weeks 0, 4, 8 and 12. VHI analyzes the following five components on a scale of 1 to 5: elasticity, fluid volume, pH, epithelial integrity, and moisture.A minimal total score of 5 points indicates severe VVA, and a maximal total score of 25 points indicates no clinical signs of VVA
improvement in Vulvovaginal atrophy (VVA) symptoms using the Visual analog scale (VAS). | 12 week
  Vulvovaginal atrophy (VVA) will be assessed at weeks 0, 4, 8 and 12. Participants will report intensity of VVA symptoms using a 10-cm VAS. The scale's left extremity indicates the complete absence of symptoms (0) and the right extremity indicates the worst possible symptom (10). Participants rated VVA symptoms (dyspareunia, dryness, or burning) from 0 to 10.
Assessment of quality of sexual function using the validated Portuguese version of the Female Sexual Function Index (FSFI) | 12 week
  The FSFI will be assessed at weeks 0,4 ,8 and 12 BY FSFI questionnaire addresses six different domains (desire, arousal, lubrication, orgasm, satisfaction, and pain/ discomfort) ranging from 0 (no sexual activity in the past 4 wk) or 1 (very dissatisfied) to 5 (very satisfied). Full scale scores ranging from 2.0 (severe dysfunction) to 36.0 (absence of dysfunction) will be used to evaluate sexual function throughout the study, with increased FSFI scores correlating to an improvement of symptoms. An optimal cut score of 26, reported by Wiegel etal, is currently used to differentiate between women with and without sexual dysfunction.

SECONDARY OUTCOMES:
Assessment of tolerability and safety of Platelet rich plasma (PRP). | 12 weeks
  it is measured by the rate of "dropouts", or patients that forfeit participation in a study due to adverse effects (pain during application of the medication, vaginal infection, haematoma formation at site of injection, vaginal spotting, vaginal leakage of the medication and need to use sanitary towels to clean leakage
Assessment of tolerability and safety of estrogen vaginal cream | 12 weeks
  it is measured by the rate of "dropouts", or patients that forfeit participation in a study due to adverse effects (pain during application of the medication .vaginal spotting, vaginal leakage of the medication and need to use sanitary towels to clean leakage

CONTACTS AND LOCATIONS:
Overall Officials: rehab A aboshama, lectuer, Principal Investigator — Fayoum University
Locations (2):
- Egypt (2):
  - Fayoum university faculity of medicine, Al Fayyum, Fayoum University Zone
  - Fayoum university, Al Fayyum

IPD SHARING:
Plan to Share IPD: No